CLINICAL TRIAL: NCT03329612
Title: Remote Ischemic Preconditioning in ACS Patients
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: poor enrollment
Sponsor: Henry Ford Health System (Other)
Responsible Party: Principal Investigator, Brittany Fuller, MD, Co-Investigator, Henry Ford Health System
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: RIPC in ACS
Record Dates: First submitted 2017-10-30; First posted 2017-11-06 (Actual); Last update posted 2022-12-14 (Actual); Status verified 2022-12

CONDITIONS: Acute Coronary Syndrome; Renal Insufficiency; Ischemia, Myocardial
MeSH Terms: conditions — Acute Coronary Syndrome; Renal Insufficiency; Myocardial Ischemia

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): This group will undergo remote ischemic preconditioning with serial inflations of the blood pressure cuff to 200 mmHg followed by deflation for reperfusion for a period of 5 minutes each for a total of 4 cycles.
  Interventions: Procedure: Remote Ischemic Preconditioning
- Control (Sham Comparator): This group will undergo serial inflations of the blood pressure cuff to 40 mmHg followed by deflation for a period of 5 minutes each for a total of 4 cycles.
  Interventions: Procedure: Remote Ischemic Preconditioning

INTERVENTIONS:
Procedure: Remote Ischemic Preconditioning — Serial inflations and deflations as detailed in the arm/group descriptions.

SUMMARY:
Remote ischemic preconditioning is a process of serial blood pressure cuff inflations and deflations that are performed prior to a procedure and have been shown in various other areas (coronary bypass surgery, vascular surgery, ST elevation myocardial infarctions) to decrease the rates of adverse events related to ischemic burden and renal injury. This procedure has not yet been studied in the population presenting with an acute coronary syndrome (ACS), even though ACS patients represent the majority of patients seen in the catheterization lab. The purpose of this study is to evaluate the efficacy of this simple and safe procedure in this particular population.

ELIGIBILITY:
Inclusion Criteria:

- Presenting with an acute coronary syndrome including non-ST elevation myocardial infarction or unstable angina on optimal medical therapy with aspirin, P2Y12 inhibitors, unfractionated heparin, statin, +/- beta blocker, +/- ace inhibitor

Exclusion Criteria:

* Presenting with ST elevation myocardial infarction
* Patients requiring circulatory support
* Need for emergent percutaneous coronary intervention
* Systemic hypotension (systolic blood pressure <90 mmHg)
* Patients in cardiogenic shock defined by requiring inotropes or vasopressors
* Patients currently on hemodialysis
* Presence of an arteriovenous dialysis fistula or graft or lymphedema in either arm
* Patients enrolled in other active cardiovascular investigational studies
* Severe comorbidities with a life expectancy of less than 6 months
* Pregnant or lactating women
* Patients unable to provide consent
* Patient taking the medication glibenclamide for treatment of diabetes

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-10-26 (Actual); Primary Completion 2018-12-30 (Actual); Study Completion 2018-12-30 (Actual)

PRIMARY OUTCOMES:
Ischemic Burden | 48-72 hours
  Assess the impact of remote ischemic preconditioning on myonecrosis following percutaneous coronary intervention by examining pre and post biomarkers

SECONDARY OUTCOMES:
Clinical Outcomes | 6 months
  Assess the effects on clinical outcomes at 6 months post initial ACS event including death, MI, stroke, revascularization and hospital readmission.
Renal Injury | 48-72 hours
  Assess the effects on post procedure renal injury

CONTACTS AND LOCATIONS:
Overall Officials: Gerald Koenig, MD, Principal Investigator — Henry Ford Health System
Locations (1):
- Henry Ford Hospital, Detroit, Michigan, United States